CLINICAL TRIAL: NCT07004660
Title: Performances of Large Language Models in Kidney Allograft Diagnostics
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Principal Investigator, Marc Raynaud, PhD, Paris Translational Research Center for Organ Transplantation
Other Study IDs: LLM_vs_Patho_001
Record Dates: First submitted 2025-05-16; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplantation
Keywords: Large language model; Banff classification; Diagnosis; Kidney transplantation; Biopsy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Necker hospital: Transplant unit from Necker hospital, France
- Saint-Louis hospital: Transplant unit from Saint-Louis hospital, France

SUMMARY:
Kidney allograft rejection diagnosis relies on the complex Banff classification, but its application is limited by variability and workload. Our group previously built a scripted automation system, though it required major expert input. This study assesses whether modern LLMs can achieve similar diagnostic performance using Banff-based prompts, without extensive manual engineering.

DETAILED DESCRIPTION:
Kidney allograft rejection remains a leading cause of allograft failure. Histological diagnosis relies on the Banff classification, a complex and evolving rule based framework. While successive Banff working groups refined the guidelines over time, daily interpretation is still hampered by inter and intra pathologist variability and growing demands on renal pathologists. This is why our group previously built a fully scripted Banff automation system. However, this system demanded years of expert curation and bespoke code before reaching acceptable accuracy. Whether modern LLMs, which show high capabilities to generate consistent and transparent reasoning at scale, can match expert pathologists without such resource intensive engineering remains unknown. The present study was therefore designed to benchmark state of the art LLMs against consensus diagnoses from senior renal pathologists on a representative series of kidney allograft biopsies, and to explore whether properly engineered prompts can translate Banff rules into reliable, reproducible diagnostic output.

ELIGIBILITY:
Inclusion Criteria:

* Kidney recipients

Exclusion Criteria:

* Combined transplant

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney recipients
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2004-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Biopsy diagnosis | The biopsy will be protocol biopsies performed at 3 months and 1 year post transplant, or for-cause biopsies performed at any time post transplant.
  The diagnosis of the biopsy will be based on the latest Banff classification (2022). The diagnoses will include i) biopsies with nonspecific lesions or clean (n=40), ii) biopsies with antibody-mediated rejection (AMR) (n=40) among which 14 had acute AMR, 13 chronic active AMR and 13 chronic inactive AMR, iii) biopsies with T cell-mediated rejection (TCMR) (n=40), among which 20 had acute TCMR and 20 had chronic active TCMR, iv) biopsies with borderline for acute TCMR (n=40), v) biopsies with mixed rejection (n=40), and vi) biopsies with microvascular inflammation (MVI) (n=40) among which 20 had probable AMR and 20 had MVI without DSA and without C4d.

IPD SHARING:
Plan to Share IPD: Undecided